CLINICAL TRIAL: NCT02402803
Title: Dried Blood Spot- Statin Pilot Study
Acronym: DBS
Status: Terminated | Type: Observational
Why Stopped: No recruitment
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Noel Bairey Merz, Principal Investigator, Cedars-Sinai Medical Center
Other Study IDs: Pro00037026
Record Dates: First submitted 2015-03-25; First posted 2015-03-30 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Hyperlipidemias; Cardiovascular Diseases
MeSH Terms: conditions — Hyperlipidemias; Cardiovascular Diseases | interventions — Dried Blood Spot Testing; Phlebotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — cholesterol panel (total cholesterol, LDL-C, triglycerides, HDL-C), Apo A-I, Apo B, Apo E, IgM, plasminogen, TIMP-1, Von Willebrand factor, antithrombin III, cystatin C, mesothelin, C-reactive protein, SAA, LPS-binding protein, mannose-binding lectin, myeloperoxidase, fibrinogen, alpha-1-acid glycoprotein, soluble transferrin receptor, haptoglobin.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Dried blood spot testing and phlebotomy — At baseline and 4-6 week follow-up, a phlebotomy serum sample (5 ml) will be collected in one golden-top tube for clinical laboratory measurement of cholesterol (total cholesterol, LDL-C, triglycerides, HDL-C) . During the same phlebotomy, a fingerprick dried blood spot (DBS) sample and two lavender EDTA plasma tubes (5 ml each) will be collected for analysis of CVD protein markers

SUMMARY:
Cardiovascular disease (CVD) is the number one cause of mortality for men and women in the United States. Dyslipidemia, particularly a high low-density-lipoprotein cholesterol (LDL-C) level, is a well-established cardiovascular risk factor and the current American Heart Association guideline for CVD risk assessment recommends a lipid panel to be checked. In addition, guidelines recommend statin therapy in all patients with clinical atherosclerotic CVD, all patients with LDL-C = 190 mg/dL, patients age 40-75 years with diabetes and LDL-C 70-189 mg/dL, and patients with an estimated 10-year atherosclerotic CVD risk = 7.5%. For all of these patients, a fasting lipid panel should be drawn prior to statin initiation as well as during follow-up to assess medication and lifestyle adherence. These fasting lipid panels are obtained via conventional phlebotomy via venopuncture in an office-based or hospital laboratory setting. However, research protein quantitation with mass spectrometry and enzyme-linked immunosorbent assay (ELISA) are technologies that allow for sensitive quantitation of protein biomarkers and targets, including lipoproteins. Most importantly, multiple reaction monitoring (MRM) mass spectrometry is able to assess samples from a dried blood spot (DBS), whose advantages include minimal volume requirements, ease of sample attainment by finger stick with minimal training required, ease of transport, and sample stability.

The purpose of the proposed analysis is to 1) measure changes in CVD biomarkers before and after initiation of statin therapy and 2) compare lipid measurements by conventional phlebotomy blood samples to research protein quantitation measurements in DBS and plasma.

DETAILED DESCRIPTION:
Despite reductions in cardiovascular disease (CVD) mortality in the past 20 years, CVD remains the leading cause of mortality in the United States, accounting for ~1 of every 3 deaths. CVD costs the U.S. over $100 billion annually and is an important field for targeted primary and secondary prevention. Dyslipidemia, particularly a high low-density-lipoprotein cholesterol (LDL-C) level, is a well-established cardiovascular risk factor, and fasting lipid panels (including total cholesterol, LDL-C, triglycerides, and high-density-lipoprotein cholesterol [HDL-C]) are included in the recent 2013 ACC/AHA Risk Assessment Guidelines. Clinical trials have shown that low density lipoprotein cholesterol (LDL-C) reduction with statin therapy predicts cardiovascular event reduction. About a quarter of all adults >45 years old were on statin therapy in 2008, and this will likely increase due to the recent 2013 ACC/AHA Cholesterol Management guidelines. These guidelines recommend statin therapy in all patients with clinical atherosclerotic CVD, all patients with LDL-C = 190 mg/dL, patients age 40-75 years with diabetes and LDL-C 70-189 mg/dL, and patients with an estimated 10-year atherosclerotic CVD risk = 7.5%. For all of these patients, a fasting lipid panel should be drawn prior to statin initiation as well as during follow-up to assess medication and lifestyle adherence. These fasting lipid panels are obtained via conventional phlebotomy via venopuncture in an office-based or hospital laboratory setting.

Research protein quantitation with mass spectrometry and enzyme-linked immunosorbent assay (ELISA) are technologies that allow for sensitive quantitation of protein biomarkers and targets, including lipoproteins. Most importantly, multiple reaction monitoring (MRM) mass spectrometry is able to assess samples from a dried blood spot (DBS), whose advantages include minimal volume requirements, ease of sample attainment by finger stick with minimal training required, ease of transport, and sample stability. DBS sampling has been used for clinical and pre-clinical studies, simplifying sample collection and handling. However, research protein quantitation with mass spectrometry and ELISA has not been compared against conventional blood sample for evaluating changes in cholesterol levels during statin therapy.

While LDL-C is well-established in predicting CVD event reduction, other laboratory lipid, thrombotic and inflammatory biomarkers have been shown to be associated with atherosclerotic plaque development or CVD risk. These include Apo A-I, Apo B, Apo E, IgM, plasminogen, TIMP-1, Von Willebrand factor, antithrombin III, cystatin C, mesothelin, C-reactive protein, SAA, LPS-binding protein, mannose-binding lectin, myeloperoxidase, fibrinogen, alpha-1-acid glycoprotein, soluble transferrin receptor, haptoglobin. All of these CVD protein biomarkers can be measured by research protein quantitation techniques.

In a pilot study of 20 subjects, we aim to:

1. measure changes in a panel of CVD protein biomarkers before and after initiation of statin therapy.
2. compare clinical laboratory measurements of LDL-C and HDL-C in conventional phlebotomy blood samples with research protein quantitation mass spectrometry and ELISA measurements of LDL-C (Apo B) and HDL-C (Apo A-I) proteins in DBS and plasma.

ELIGIBILITY:
Inclusion criteria:

1. Men and women age> 18 years who are initiated on statin therapy in the clinical setting.

Exclusion criteria:

1. History of rhabdomyolysis
2. History of prior allergic reaction to statins
3. History of liver failure
4. Contraindications to antecubital phlebotomy or finger stick (including those with bilateral dialysis AV fistulae).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women age> 18 years who are initiated on statin therapy in the clinical setting
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-10; Primary Completion 2020-10 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Clinical lipid and research protein measurements (composite) | up to 4-6 week follow-up
  Compare LDL-C and HDL-C clinical laboratory test measurements in serum vs Apo B and ApoA-I research protein measurements in DBS and plasma as to correlation coefficient across subject samples and level of response (expected reduction) in LDL/Apo B following initiation of statin therapy

SECONDARY OUTCOMES:
Biomarker change | Baseline and 4-6 week follow-up
  Compare biomarker changes Pre- vs Post-statin treatment as observed by LDL-C and HDL-C clinical laboratory tests, research protein measurements in plasma and in dried blood spot
Research protein measurements in dried blood spot vs plasma | Baseline and 4-6 week follow-up
  3) Compare research protein measurements of CVD protein markers in dried blood spot and plasma samples to investigate parallelism of results
Clinical Cardiovascular Risk Score | Baseline
  Compare the research protein measurements of CVD protein markers with the ACC/AHA 10-year atherosclerotic CVD risk score

CONTACTS AND LOCATIONS:
Overall Officials: C. Noel Bairey Merz, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes